CLINICAL TRIAL: NCT01244867
Title: A Phase 2, Randomized, Observer-blind, Single Center, Dose-Ranging Study to Evaluate the Immunogenicity Safety and Tolerability of the H5 VLP Influenza Vaccine With or Without Alhydrogel in Healthy Adults 18-60 Years of Age.
Brief Title: Immunogenicity, Safety, Tolerability of a Plant-Made H5 VLP Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-H5VLP-002
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 20 microgram H5 VLP vaccine + Alhydrogel (Experimental)
  Interventions: Biological: 20 micrograms dose H5 VLP
- 30 micrograms H5 VLP vaccine + Alhydrogel (Experimental)
  Interventions: Biological: 30 micrograms dose H5 VLP
- 45 micrograms H5 VLP vaccine + Alhydrogel (Experimental)
  Interventions: Biological: 45 micrograms dose H5 VLP
- 45 micrograms H5 VLP vaccine (Experimental)
  Interventions: Biological: 45 micrograms non-adjuvanted H5 VLP
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 20 micrograms dose H5 VLP — 2 doses given 21 days apart of 20 micrograms of H5 VLP vaccine mixed with Alhydrogel
  Arms: 20 microgram H5 VLP vaccine + Alhydrogel
Biological: 30 micrograms dose H5 VLP — 2 doses given 21 days apart of 30 micrograms of H5 VLP vaccine mixed with Alhydrogel
  Arms: 30 micrograms H5 VLP vaccine + Alhydrogel
Biological: 45 micrograms dose H5 VLP — 2 doses given 21 days apart of 45 micrograms of H5 VLP vaccine mixed with Alhydrogel
  Arms: 45 micrograms H5 VLP vaccine + Alhydrogel
Biological: 45 micrograms non-adjuvanted H5 VLP — 2 doses given 21 days apart of 45 micrograms of H5 VLP vaccine
  Arms: 45 micrograms H5 VLP vaccine
Biological: Placebo — 2 doses given 21 days apart of the placebo
  Arms: Placebo

SUMMARY:
The primary objective is to assess the immunogenicity and safety and tolerability of two consecutive doses of H5 VLP Influenza vaccine given 21 days apart, at three dose levels: in part A: 20 µg, 30 µg and 45 µg combined with Alhydrogel® 1%, or 45 µg without Alhydrogel®, compared to the placebo, (100mM phosphate buffer + 150mM NaCl + 0.01% Tween 80).

DETAILED DESCRIPTION:
An adaptive design is proposed for this phase 2 trial. Part A of this study will consist of dose-ranging in 135 subjects who will be randomized to receive one injection of either 20 µg, 30 µg or 45 µg H5 VLP Influenza vaccine combined with Alhydrogel®, or 45 µg without Alhydrogel®, or the placebo preparation, (100mM phosphate buffer + 150mM NaCl + 0.01% Tween 80) at Days 0 and 21. Seven-day (7) safety data after the first immunization for subjects in all five treatment groups will be tabulated and reviewed by a panel consisting of 2 external medical advisors, prior to permitting the second immunization of vaccine/placebo for all treatment groups at Day 21 (Part A). Twenty-one (21) days after the last subject vaccine administration in Part A, all safety and immunogenicity data will be collected and analysed to determine the optimal dose level. Following selection of the optimal dose, Part B of the trial will commence and consist of administration of the selected optimal dose(s) in one hundred (100) subjects, plus administration of placebo in twenty (20) subjects (total of 120 subjects in part B). These subjects will similarly receive two vaccinations 21 days apart and will be followed in the exact same fashion as Part A, except that there will be no 7-day safety analysis. Depending on data analysis one or a maximum of two vaccine doses could be selected to be further evaluated during part B of the trial. All Part A and B subjects will be followed for safety until Day 228.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 to 60 years of age;
* Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, vital signs, screening laboratories and medical history conducted no more than 30 days prior to study vaccine administration;
* BMI of ≥18 and ≤ 32;
* Comprehension of the study requirements, expressed availability for the required study period and ability to attend scheduled visits;
* Accessible by telephone on a consistent basis;
* In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee;
* If female and capable of child-bearing, have a negative serum pregnancy test result at study entry, has been consistently using effective birth control for the 28 days prior to study entry and agree to continue employing adequate birth control measures for the duration of the study.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

  1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
  2. Requiring a change in medication dosage in one month prior to test article administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  3. Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to test article administration;
* Any medical or neuropsychiatric condition which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting;
* Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection or Hepatitis B or C or presence of lymphoproliferative disease;
* Presence of any febrile illness, oral temperature of >38.0˚C within 24 hours of test article administration. Such subjects may be re-evaluated for enrolment after resolution of illness;
* History of autoimmune disease;
* Administration of any vaccine (including any other influenza vaccine) within a 30 day period prior to study enrolment, or planned administration within the period from the first vaccination up to blood sampling at Day 42 or within 30 days prior to blood sampling at Day 228. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to test article administration. Receipt of any other emergency immunizations (e.g. rabies) will result in a case-by-case review of continued participation;
* Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other drug study while participating in this study;
* Treatment with systemic glucocorticoids at a dose exceeding ≥ 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of first test article administration, or any other cytotoxic or immunosuppressant drug or any immune globulin preparation within three months of vaccination. Nasal or inhaled glucocorticoids are allowed;
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin, and without a clinically apparent bleeding tendency are eligible;
* History of previous H5N1 vaccination or a history of exposure to H5N1 virus;
* History of allergy to any of the constituents of H5 VLP (H5N1) study vaccine, Alhydrogel® (aluminum hydroxide), or the phosphate buffer;
* History of severe allergic reactions or anaphylaxis;
* History of tobacco allergy;
* History of anti-histaminics used continuously for 4 weeks or more at any time in the past year;
* Have a rash, dermatological condition or tattoos which may interfere with injection site reaction rating;
* Have received a blood transfusion or immunoglobulins within 90 days of study entry;
* If female, and of childbearing potential, has not been consistently using effective birth control for the 28 days prior to study entry. An example of highly effective birth control is oral contraceptives, hormone implants, abstinence (confirmed by Investigator), or male condom plus spermicide. All female subjects, regardless of birth control history must provide a serum sample for pregnancy screening. Effective birth control must be used for the duration of the study for female of child bearing potential must have no plan to become pregnant during the study period.;
* Among female subjects, either known pregnancy or urine beta-human chorionic gonadotropin (ß-hCG) test results consistent with pregnancy prior to test article administration on Day 0;
* Female subjects who are lactating;
* Vital sign abnormalities: systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥90 mmHg, resting pulse rate <40 bpm or >100 bpm or according to the Investigator's opinion;
* Cancer or treatment for cancer within 3 years of test article administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 21 days after each injection and 6-month follow-up period
  Immunogenicity Geometric mean titres: (GMTs) of hemagglutination inhibition (HI) antibody on Days 0, 21 and 42. Follow-up serology samples for GMTs will be taken at Day 228.
Safety | 21 days after each vaccination and 6-month follow-up
  Safety will be assessed by the rate and severity of solicited and unsolicited adverse events post-vaccination. A 6-month follow-up period will be performed.

SECONDARY OUTCOMES:
Immunogenicity | 21 dyas after each injection
  The secondary objective is to assess the cross-reactivity of antibodies induced by two consecutive doses of H5 VLP influenza vaccine given 21 days apart, at three dose levels: 20 µg, 30 µg and 45 µg combined with Alhydrogel® 1%, or 45 µg without Alhydrogel® 1% as measured by HI antibody titers for the A/Vietnam/1203/04, A/Anhui/01/2005 and A/turkey/Turkey/1/05 H5N1 strains and as measured by MicroNeutralisation(MN) antibody titers for the A/Indonesia/5/05 and A/Vietnam/1203/04 H5N1 strains.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M. Sellers, MD, Principal Investigator — Kendle Early Stage Toronto Canada
Locations (1):
- Kendle Early Stage, Toronto, Ontario, Canada